CLINICAL TRIAL: NCT05866887
Title: Insomnia Prevention in Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric Zhou, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-677; R03CA259894-01 (NIH)
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Acute Lymphoblastic Leukemia; Leukemia; Acute Lymphoblastic Leukemia
Keywords: Pediatric Acute Lymphoblastic Leukemia; Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep ALL Night (Experimental): Participants and parents will complete study procedures as outlined:
  * Baseline survey completed by participant parent(s).
  * Introduction to Sleep ALL Night action plan.
  * Review of psychoeducational website and completion of sleep diary.
  * Survey completed by participant parent(s).
  Interventions: Behavioral: Sleep ALL Night

INTERVENTIONS:
Behavioral: Sleep ALL Night — Sleep intervention program comprised of a sleep action plan tool and interactive psychoeducation website.

SUMMARY:
The goal of this research study is to understand the acceptability and feasibility of the Sleep ALL Night intervention among children with Acute Lymphoblastic Leukemia (ALL) in hopes of improving the discussion of sleep disorders with clinical providers.

The name of the intervention used in this research study is: Sleep ALL Night, which is a sleep intervention program comprised of an action plan tool and psychoeducational website.

DETAILED DESCRIPTION:
This research study is to conduct a single-arm pilot study to determine the acceptability and feasibility of Sleep ALL Night for children with Acute Lymphoblastic Leukemia (ALL).

Participation in this research study is expected to last 1 month.

It is expected about 30 children will take part in this research study.

The National Cancer Institute (NCI) is providing funding for this research study through a grant.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the Maintenance Phase of therapy on or as per DFCI 16-001 and has completed at least two cycles of maintenance therapy to allow adequate recovery from the more intensive Consolidation phase.
* English or Spanish speaking child and primary caregiver (parent/guardian).
* Child aged 4-12 years.

Exclusion Criteria:

* Primary team declines permission to approach.
* Children with critical illness (defined as ICU admission)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Zhou, PhD, Principal Investigator — Dana-Farber Cancer Institute; Kira Bona, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sleep ALL Night: Single-arm study where participants receive a single meeting to discuss and review study materials regarding sleep health in pediatric ALL patients.
Period: Overall Study
Arm/Group | Sleep ALL Night
Started | 25
Completed | 22
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sleep ALL Night
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.6 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate of Participants
Description: The primary study outcome of acceptability is defined as the proportion of eligible participants who are approached by research staff who agree to participate in the study, with the cutoff set at ≥30% of eligible participants who are approached agreeing to participate.
Time Frame: At screening, when eligible participants are approached by research staff. Recruitment occurred over a 5-month period.
Population: The number of participants analyzed (27) is greater than the number enrolled on the study (25) because not all participants were either eligible or interested in study enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep ALL Night
Number analyzed (Participants) | 27
Participants | 25

2. Primary Outcome: Acceptability of Intervention Measure Scale Score
Description: The primary study outcome of acceptability is defined as participants reporting an average score of ≥4 ("Agree") on the Acceptability of Intervention Measure scale, a four-item questionnaire assessing the acceptability of an intervention. The scale uses a 5-point scale with options ranging from Completely Agree (5) to Completely Disagree (1). The average score of all four items was used as the primary outcome. A higher score indicates greater belief that the intervention was acceptable for the participant.
Time Frame: At Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep ALL Night
Number analyzed (Participants) | 22
score on a scale | 4.40 (0.63)

3. Primary Outcome: Intervention Assessment Completion Rate
Description: The primary study outcome of feasibility is defined as ≥80% of enrolled participants complete the Post-Intervention Assessment.
Time Frame: Up to 1 month after the conclusion of the study period, up to 8 weeks.
Population: Number of participants who completed the Post-Intervention Assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep ALL Night
Number analyzed (Participants) | 25
Participants | 22

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Sleep ALL Night
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
Feasibility and acceptability trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT05866887/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT05866887/ICF_001.pdf